CLINICAL TRIAL: NCT06030661
Title: The HF-POL Study - Multicenter Study of Polish Patients With Heart Failure and Left Ventricular Ejection Fraction >40%
Brief Title: The HF-POL Study - Multicenter Study of Polish Patients With HF and LVEF >40%
Acronym: HF-POL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Lodz (Other)
Collaborators: Medical University of Silesia (Other); University of Opole (Other); Medical University of Warsaw (Other); Wroclaw Medical University (Other); Military Institute od Medicine National Research Institute (Other); Jagiellonian University (Other); Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland (Other); Medical University of Bialystok (Other); Świętokrzyskie Cardiology Center of Kielce (Unknown); Regional Specialist Hospital in Rybnik (Unknown)
Responsible Party: Sponsor
Other Study IDs: RNN/240/21/KE
Record Dates: First submitted 2023-08-30; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Heart Failure
Keywords: heart failure with preserved ejection fraction; heart failure with mildly reduced ejection fraction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
HF-POL is the first Polish multicenter observational prospective registry of patients with heart failure and ejection fraction more than 40% designed by Heart Failure Association of the Polish Cardiac Society. The purpose of this study was to provide first characteristics of Polish population patients with heart failure and EF>40% and to provide a better understanding of medical practice, based on observational data, including diagnosis, treatment, and prognosis over 3-year follow-up.

DETAILED DESCRIPTION:
HF-POL is the first Polish multicenter observational prospective registry of patients with heart failure and ejection fraction more than 40%. HF-POL study is conducted by the Heart Failure Association of the Polish Cardiac Society in cooperation with the Committee for Clinical Initiatives of the Executive Board as part of the Scientific Platform initiative. The leading center of the study is the Military Medical Academy Memorial Teaching Hospital of the Medical University of Lodz, Poland. The Primary Investigator is Malgorzata Lelonek; the Steering Committee includes Malgorzata Lelonek, Mariusz Gasior, and Marcin Grabowski. The study was approved by the Bioethics Committee at the Medical University of Lodz (No. RNN/240/21/KE; October 21, 2021).

The purpose of this study was to provide first characteristics of Polish population patients with heart failure and EF>40% and to provide a better understanding of medical practice, based on observational data, including diagnosis, treatment, and prognosis over 3-year follow-up. Patients have been recruited at each participating center since that center's activation on the eCRF.biz platform (a clinical data management system, https://rejestr.gbbsoft.pl/hf-pol). We collected data included demographics, medical history, concomitant medications, selected laboratory, electrocardiographic and echocardiographic results as well ascomorbidities. Patients are diagnosed and treated according to the current clinical practice guidelines and the standard of care at participating centers.

All consecutive patients meeting the inclusion and exclusion criteria are being enrolled.

Heart Failure should be recognized according to the 2021 ESC guidelines. The study allows recruitment based on results from medical records, especially for outpatients with a history of Heart Failure. The study population includes patients with Heart Failure and LVEF >40%. In total, a minimum of 1000 patients from 14 Polish centers will be enrolled.

Patients will stay in 3-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* documented EF >40%
* symptomatic chronic Heart Failure or acute Heart Failure (worsening of chronic Heart Failure or Heart Failure de novo) requiring hospitalization and intravenous agents

Exclusion Criteria:

* age <18 years
* dyspnea due to other causes than Heart Failure.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Polish population with Heart Failure and EF >40%.
Sampling Method: Non-Probability Sample
Enrollment: 1497 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Death andr/or the first heart failure hospitalisation | From randomisation to end-of-study ( 3 years)
  Occurrence of all-cause mortality and/or the first heart failure hospitalisation

SECONDARY OUTCOMES:
All heart failure hospitalisations | From randomisation to end-of-study (3 years)
  Number of heart failure hospitalisations
All cause hospitalisations | From randomisation to end-of-study ( 3 years)
  Number of all cause hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Lelonek, Prof.MD, PhD, Principal Investigator — Medical University of Lodz
Locations (1):
- Department of Noninvasive Cardiology, Medical University of Lodz, Lodz, Poland